CLINICAL TRIAL: NCT07367607
Title: Circadian Modulation of Neurophysiological Responses to Therapeutic Massage Modalities in Taekwondo Athletes: A Randomized Crossover Trial
Brief Title: Circadian Modulation of Neurophysiological Responses to Therapeutic Massage Modalities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Princess Nourah Bint Abdulrahman University (Other)
Responsible Party: Principal Investigator, Monira Aldhahi, Associate Prof, Princess Nourah Bint Abdulrahman University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PNU-10
Record Dates: First submitted 2026-01-17; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Healthy
MeSH Terms: interventions — N-formylmethionylphenylalanine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Friction Massage (FMP) (Experimental)
  Interventions: Behavioral: FMP
- Vibration Mechanical Massage (VMMP) (Experimental)
  Interventions: Device: VMMP
- Percussion Mechanical Massage (PMMP) (Experimental)
  Interventions: Device: PMMP

INTERVENTIONS:
Behavioral: FMP — Manual therapeutic massage consisting of rhythmic, sustained friction techniques applied by a certified physiotherapist to the dominant upper extremity muscles. Moderate-to-strong pressure was applied for a total duration of 10 minutes using a standardized intermittent protocol.
  Arms: Friction Massage (FMP)
Device: VMMP — Therapeutic vibration massage delivered using a handheld vibration device set at a fixed frequency of 50 Hz. The device was applied to the dominant upper extremity muscles for 10 minutes to provide localized high-frequency mechanical stimulation.
  Arms: Vibration Mechanical Massage (VMMP)
Device: PMMP — Therapeutic percussion massage administered using a handheld percussive therapy device delivering rapid mechanical impulses at approximately 40 Hz. The intervention was applied to the dominant upper extremity muscles for 10 minutes to elicit deep somatosensory stimulation.
  Arms: Percussion Mechanical Massage (PMMP)

SUMMARY:
Athletic performance and recovery are closely linked to central nervous system regulation, which can be objectively assessed using electroencephalography (EEG). Although therapeutic massage is widely used as a recovery modality in combat sports, its neurophysiological effects and potential interaction with circadian timing remain poorly understood. This study investigates whether different therapeutic massage modalities applied at different times of the day modulate resting-state EEG activity in taekwondo athletes.

DETAILED DESCRIPTION:
This randomized, within-subject crossover study examines the effects of different therapeutic massage modalities and time of day on resting-state EEG activity in elite male taekwondo athletes. Twelve athletes complete four experimental conditions: no-massage control, friction massage, vibration mechanical massage, and percussion mechanical massage. Each condition is administered during both morning and evening sessions, separated by a minimum 48-hour washout period.

Resting-state EEG is recorded immediately following each intervention using a 32-channel system. Power spectral density is computed to extract global band power in delta, theta, alpha, beta, and gamma frequency bands. The study aims to determine whether massage modality, circadian timing, or their interaction significantly influences cortical oscillatory activity associated with recovery and neural readiness.

ELIGIBILITY:
Inclusion Criteria:

* Male taekwondo athletes aged 18-25 years
* Minimum of 4 years of structured taekwondo training
* Training frequency ≥ 5 days/week
* Black belt (1st Dan or higher)
* No musculoskeletal injury in the past 6 months

Exclusion Criteria:

* Neurological or psychiatric disorders
* Use of stimulant substances or anti-inflammatory medication
* Irregular sleep-wake patterns (e.g., shift work)
* Withdrawal of consent at any stage

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-01-05 (Actual)

PRIMARY OUTCOMES:
Global EEG Band Power | Immediately post-intervention in morning and evening sessions.
  Log-transformed power spectral density values for delta, theta, alpha, beta, and gamma frequency bands obtained from resting-state EEG recordings.

SECONDARY OUTCOMES:
Topographical EEG Distribution | Immediately post-intervention in morning and evening sessions.
  Spatial distribution of EEG band power across frontal and central scalp regions.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Sport Sciences, İnönü University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided